CLINICAL TRIAL: NCT04716920
Title: Tai Chi for Relieving Aromatase Inhibitor-Induced Arthralgia in Breast Cancer Patients
Brief Title: Tai Chi for Relieving Aromatase Inhibitor-Induced Arthralgia in Patients With Stage I-III Breast Cancer, the TaiChi4Joint Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20G.093; NCI-2020-02555 (Other: The Buck Foundation); JT 14910 (Other: JeffTrial Number)
Record Dates: First submitted 2020-12-07; First posted 2021-01-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Tai Chi, Fitbit, Tai4Chijoint group) (Experimental): Patients attend Tai Chi exercise classes over 1 hour BIW and wear a Fitbit device for up to 12 weeks. Patients are encouraged to complete self-practice over 30 minutes and record practice times daily in a diary log form. Patients also join a Facebook private TaiChi4joint group where they receive instructional videos matching the progress of weekly classes for at-home practices and peer support in Tai Chi engagement.
  Interventions: Other: Tai Chi; Device: FitBit; Other: Support Group Therapy; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Tai Chi — Attend Tai Chi exercise classes
Device: FitBit — Wear FitBit
Other: Support Group Therapy — Join Tai4Chijoint group
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This trial studies new methods using Tai Chi for the relief of joint pain (arthralgia) caused by an aromatase inhibitor in patients with stage I-III breast cancer. Tai Chi is a mind-body therapy that integrates moderate physical activity, deep breathing and meditation. Tai Chi may help to reduce aromatase inhibitor-induced joint pain, and offer a promising approach to managing symptoms in cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility, acceptability, and preliminary efficacy of a 12-week Tai Chi intervention for relieving aromatase inhibitor (AI)-induced arthralgia in women with breast cancer (BCa).

OUTLINE:

Patients attend Tai Chi exercise classes over 1 hour twice weekly (BIW) and wear a Fitbit device for up to 12 weeks. Patients are encouraged to complete self-practice over 30 minutes and record practice times daily in a diary log form. Patients also join a Facebook private TaiChi4joint group where they receive instructional videos matching the progress of weekly classes for at-home practices and peer support in Tai Chi engagement.

ELIGIBILITY:
Inclusion Criteria:

* Be able to speak and read English
* Been diagnosed with stage I-III breast cancer (BC)
* Had completed all active treatments
* Had been receiving an AI (anastrozole, letrozole, or exemestane) for at least 3 months
* Had joint (knee, hand or hip) pain or stiffness that started or worsened after the initiation of AI
* Report worst pain in the past week >= 4 on a 0-10 numeric rating scale
* Be willing to adhere to all study procedures

Exclusion Criteria:

* Has been diagnosed with another form of cancer in the past 5 years
* Uncontrolled cardiac, pulmonary, or infectious disease
* Body mass index (BMI) > 40 kg/m^2
* Currently attending any mind-body therapy classes (e.g. yoga)
* Joint pain due to inflammatory arthritic condition (such as rheumatoid arthritis, osteoarthritis or gout, which will be assessed during eligibility screening with patient self-reported data and will be screened through electronic medical record [EMR] data)
* Had surgery or joint infection in the past 6 months
* Currently taking corticosteroids or opioids, have discontinued or plan to discontinue AI in the next 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Tai Chi practice | Up to 12 weeks
  Diary log form.
Tai Chi practice | Up to 12 weeks
  Examples include documenting potential issues that participants think might be intervention-related.
Assess the client's perspective on the value of services received | Up to 36 weeks
  Will be assessed using the Client Satisfaction Questionnaire. Qualitatively, five questions, adapted from previous yoga research will be used in post-intervention patient interview.
Lower-extremity joint symptoms | Up to 12 weeks
  Western Ontario and McMaster Universities Arthritis Index will be used to assess pain in the past 7 days in three domains: pain, stiffness, and physical function; higher scores indicating worse pain, stiffness, and functional limitations.
Pain, stiffness, and physical function in the hands | Up to 12 weeks
  Australian/Canadian Osteoarthritis (OA) Hand Index will be used to assess pain, stiffness, and physical function in the hands.
Assess pain, pain severity, and pain interference | up to 12 weeks
  Brief Pain Inventory will be used to assess worst pain, pain severity, and pain interference over the past week.
Fatigue | Up to 12 weeks
  Fatigue Symptom Inventory will be used to measure change in fatigue among breast cancer (BCa) patients and with strong internal consistency.
Effects of Hot Flashes on Quality of life | Up to 12 weeks
  Hot Flash Related Daily Interference Scale will be used to measure the effect of hot flashes on overall quality of life and on nine specific activities: work, social activities, leisure activities, sleep, mood, concentration, relations with others, sexuality, and enjoyment of life.
Assessment of Sleep quality | Up to 12 weeks
  Pittsburg Sleep Quality Index will be used to for subjective sleep assessment, which includes multiple sleep-related variables over the preceding month.
Cancer-related distress | Up to 12 weeks
  Centers for Epidemiologic Studies Depression Scale will be used to assess depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gomaa S, West C, Lopez AM, Zhan T, Schnoll M, Abu-Khalaf M, Newberg A, Wen KY. A Telehealth-Delivered Tai Chi Intervention (TaiChi4Joint) for Managing Aromatase Inhibitor-Induced Arthralgia in Patients With Breast Cancer During COVID-19: Longitudinal Pilot Study. JMIR Form Res. 2022 Jun 21;6(6):e34995. doi: 10.2196/34995. PMID 35727609